CLINICAL TRIAL: NCT04867005
Title: Measuring the Effectiveness of a Training Program for the Implementation of Advance Care Planning in Primary Care Teams: a Cluster Randomized Clinical Trial
Brief Title: Advance Care Planning in Primary Care: a Cluster Randomized Clinical Trial
Acronym: PDA_CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Cristina Lasmarias, PhD, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PDA001
Record Dates: First submitted 2021-04-19; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Self Efficacy
Keywords: Advance Care Planning; Cluster Randomized clinical trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online traininig group. A (Active Comparator): This arm included 5 primary care teams, that carried out a 10 hours online course.
  Interventions: Behavioral: Impact of a training program
- online and face-to-face training group. B (Experimental): This arm included 5 primary care teams, that carried out a 10 hours online course plus a 6h hours face-to-face course
  Interventions: Behavioral: Impact of a training program

INTERVENTIONS:
Behavioral: Impact of a training program — Measurement of the effectiveness of a training program based on the skills and knowledge learning on advance care planning. A 10 hours online course was administered to both arms through an online platform; the 6 hours face-to-face course was administered to each primary care team (5) included in this arm. The 6 hours course was split into 2 sessions of 3 hours each.
  Other Names: Self-efficacy improvement on Advance Care Planning

SUMMARY:
The study on the effectiveness of a training program in Advance Care Planning (ACP) with primary care professionals has been designed as a cluster-randomized clinical trial.

Aim: To measure the effectiveness of a training program on ACP in Primary healthcare professionals in a population area of Catalonia. Design: Cluster Randomized clinical trial with a measure of pre-post effectiveness between groups of intervention based on the measurement of self-efficacy in advance care planning. Scope: Barcelona Nord and Maresme (BNM). Population: Primary care doctors and nurses. Sample: doctors and nurses from the Primary Care Service (SAP) of the BNM. The study is divided into 3 phases: 1) Planning: training design, randomization and parallel assignment in 2 arms, online training versus online and face-to-face training; 2) Implementation: data collection pre-intervention and training; 3) Evaluation: post data collection (1 follow-up 4 months after recruitment/ after training) and data analysis. Intervention: both arms (A and B) will carry out the online training which consists of a 10 hours course. Arm B will also do the 6-hour face-to-face workshop, divided into two sessions of 3 hours. Primary outcome: ACP Self-efficacy (using a validated scale Advance Care Planning-Self Efficacy Spanish (ACP_SEs). Secondary outcomes: Socio-demographic: age, gender, years of professional experience and in the professional field, previous knowledge in ACP, previous training in ACP; training Satisfaction; ACP Registration Variables in the medical records of patients identified as chronic advanced patients:% clinical records with ACP processes registration, identification of the surrogate decision-maker, values, preferences, and specific decisions records, identification of the place of care and of death preferred, adequacy of the place of death in case of death. Analysis: calculation of the sample applying correction values for the cluster effect; mean, median, range, confidence interval, and standard deviation of quantitative variables and absolute and relative frequency of qualitative variables. Pre- and post-comparison for the measurement of variance (ANOVA) resulting between the intervention groups from the chi-square test; multivariate logistic regression model and 5% significance level

ELIGIBILITY:
Inclusion Criteria:

* Cluster inclusion criteria:

  • Being a primary care team belonging to SAP BNM.
* Individuals inclusion criteria:

  * Being a doctor or a nurse working at the primary care teams recruited.
  * 280 will take part in the study, belonging to the 10 primary care teams recruited.

Exclusion Criteria:

* Cluster inclusion criteria:

  • Being teams that share Primary Care Center, in order to avoid contamination between clusters as long as they share patient assignment.
* Individuals inclusion criteria:

  * Professionals who refuse to be part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Advance care planning self-efficacy (ACP-SEs) | 4 months
  Self-efficacy on Advance care planing was measured through a recently validated scale into spanish. This scale includes 19 items and it is a 5-point likert scale (1 not at all capable/ 5 completely capable). Due to self-efficacy is a subjective item, no worse o better score is considered. Measurements were collected before training and immediately after training

SECONDARY OUTCOMES:
Clinical records on Advance care planning | 5 months
  The clinical records of advanced chronic patients were measured in order to evaluate how ACP were registered before and after the intervention
Satisfaction with the training process | 1 month
  Satisfaction was measured after training on both arms. An ad-hoc 6 point likert ad questionaire was created, including 20 items: satisfaction with contents, organization, teacher, among others...
Knowledge acquired | 4 months
  An ad-hoc 12 items test was created. This outcome was measure before and after training . Correct answers were compared

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Eap Arenys de Mar, Arenys de Mar, Barcelona
  - Eap Gatassa - Mataró 6, Mataró, Barcelona
  - Eap La Riera - Mataró-1, Mataró, Barcelona
  - Eap Rocafonda-El Palau - Mataró 3, Mataró, Barcelona
  - Eap Ronda Cerdanya - Mataró 5, Mataró, Barcelona
  - Eap Ronda Prim - Mataró 7, Mataró, Barcelona
  - Eap Premià de Mar, Premià de Mar, Barcelona
  - Eap Sant Andreu de Llavaneres, Sant Andreu de Llavaneres, Barcelona
  - Eap Vilassar de Dalt, Vilassar de Dalt, Barcelona
  - Eap Vilassar de Mar, Vilassar de Mar, Barcelona

IPD SHARING:
Plan to Share IPD: No